CLINICAL TRIAL: NCT00987181
Title: Non Contact Measurement of Aortic Pulse Wave Velocity
Brief Title: Non-Contact Measurement of Aortic Compliance
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Stephen Greenwald, Professor of Cardiovascular Mechanics, Barts & The London NHS Trust
Other Study IDs: II-FS-0109-11005; i4i Track 1
Record Dates: First submitted 2009-09-15; First posted 2009-09-30 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Vascular Disease
Keywords: Pulse wave velocity; Non contact; Non-invasive; Photoplethysmography; Doppler flow velocimetry
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Angiography high risk: Patients with multiple risk factors, positive non-invasive test, or known pre-existing coronary artery/vascular disease. Patients with diabetes mellitus will be identified, and subject to a sub-group analysis.
- Angiography Low Risk: Patients with chest pain symptoms, minimal risk factors, and inconclusive evidence of myocardial ischaemia on non-invasive testing.

SUMMARY:
Reduced aortic stiffness is a powerful way to predict the outcome of cardiovascular (CV) disease. There are several non invasive methods for its estimation, most of which are based on the measurement of speed of the arterial pulse wave. (The stiffer the artery, the faster the pulse wave travels.) They rely on detecting the arterial pulse with 2 sensors placed on the skin a known distance apart and measuring the time for the pulse to travel between them. However all current methods require skilled operators and are of limited accuracy. Thus, there is a need for an easy to use and reliable device to measure pulse speed. The aim of this project is to develop a non contact device to detect the aortic pulse as it moves into the small arteries following the ribs, using the principle of thermal imaging, by means of a high sensitivity infra red camera, directed towards the subjects back. The investigators plan to validate the device and conduct a small feasibility study in patients undergoing elective angiography, by simultaneously measuring pulse speed using established methods. These are Doppler ultrasound (non-invasive) and direct intra-arterial measurement (the gold standard).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Patients eligible for coronary angiography
* Informed consent obtained
* Able to complete experimental protocol

Exclusion Criteria:

* Refusal of consent
* Age below 18 years
* Breast feeding
* Known or suspected pregnancy
* Patient participating in another study at time of study entry or previous participation in this registry
* diagnosed but untreated hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-interventional cardiology clinic. Patients undergoing elective angiography.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-09; Primary Completion 2012-06 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Quantitative agreement between intra-arterial measurement of aortic pulse wave velocity and transcutaneous values: a) Contact PPG from probes on the skin of the back in the intercostal spaces and b) non-contact from infra-red camera imaging the back. | Single measurement to be made between January 2010 and June 2010

SECONDARY OUTCOMES:
Assessment of differences in aPWV and between low and high risk groups of patients undergoing elective coronary angiography. | Single measurement to be made between January 2010 and June 2010

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Greenwald, PhD, Principal Investigator — Queen Mary University of London, Barts & The London School of Medicine & Dentistry
Locations (1):
- London Chest Hospital, London, London, United Kingdom

REFERENCES:
- [Background] Greenwald, S.E., Denyer, H.T., and Sobeh, M.S., Non Invasive Measurement of Vascular Compliance by a Photoplethysmographic Technique. SPIE Proc., 1997. 2970: 89-97.
- [Background] Loukogeorgakis S, Dawson R, Phillips N, Martyn CN, Greenwald SE. Validation of a device to measure arterial pulse wave velocity by a photoplethysmographic method. Physiol Meas. 2002 Aug;23(3):581-96. doi: 10.1088/0967-3334/23/3/309. PMID 12214765
- [Background] Zheng, J., Hu., S., Azorin-Peris, V., Echiadis, A., Shi, P., Chouliaras, V., "A remote approach to measure blood perfusion from the human face", Vol. 7170. 7170-4., Proc. of SPIE BiOS
- [Background] Cohn JN, Duprez DA, Grandits GA. Arterial elasticity as part of a comprehensive assessment of cardiovascular risk and drug treatment. Hypertension. 2005 Jul;46(1):217-20. doi: 10.1161/01.HYP.0000165686.50890.c3. Epub 2005 May 2. PMID 15867132
- [Background] Greenwald SE. Ageing of the conduit arteries. J Pathol. 2007 Jan;211(2):157-72. doi: 10.1002/path.2101. PMID 17200940
- [Background] Mitchell, G.F., Pulse Wave Velocity Measuring Device, USA, 2001, 6331162 B1.
- [Background] Rajzer MW, Wojciechowska W, Klocek M, Palka I, Brzozowska-Kiszka M, Kawecka-Jaszcz K. Comparison of aortic pulse wave velocity measured by three techniques: Complior, SphygmoCor and Arteriograph. J Hypertens. 2008 Oct;26(10):2001-7. doi: 10.1097/HJH.0b013e32830a4a25. PMID 18806624
- [Background] Wang X, Keith JC Jr, Struthers AD, Feuerstein GZ. Assessment of arterial stiffness, a translational medicine biomarker system for evaluation of vascular risk. Cardiovasc Ther. 2008 Fall;26(3):214-23. doi: 10.1111/j.1755-5922.2008.00051.x. PMID 18786091